CLINICAL TRIAL: NCT04484922
Title: The Effect of Dexmedetomidine on Neuroprotection in Pediatric Cardiac Surgery Patients: a Randomized Controlled Trial
Brief Title: Dexmedetomidine Neuroprotection in Pediatric Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2001-062-1095
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — continuous infusion of dexmedetomidine during the surgery
  Arms: Dexmedetomidine
Drug: Normal saline — continuous infusion of normal saline during the surgery
  Arms: Control

SUMMARY:
Neurodevelopmental disability is the most significant complication for survivors of infant surgery for congenital heart disease. In this study we sought to determine if intraoperative continuous infusion of dexmedetomidine are associated with neurodevelopmental outcomes at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Neonates undergoing cardiac surgery
* Infants undergoing cardiac surgery with cardiopulmonary bypass (atrial septal defect repair, ventricular septal defect repair, or tetralogy of fallot repair)

Exclusion Criteria:

* History of hypersensitivity of any drug
* Presence of hypotension or bradycardia considering age Bradycardia (heart rate < 80 beats/min) or hypotension (systolic blood pressure < 70mmHg for infants, < 60mmHg for neonates)
* Elevated liver enzyme levels (aspartate transaminase >100unit/L, alanine aminostrasferase > 50 unit/L)
* surgery with deep hypothermic circulatory arrest
* Presence of complex cardiac defect
* single ventricular physiology
* plan of additional operation within a year
* preoperative use of beta-agonists
* presence of history of any neurological disorder

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Bayley scales of Infant development | 1 year after the surgery
  Developmental outcomes at each assessment and within each domain (cognitive, language, and motor) were classified as "average" if they were within 1 SD of the mean or higher (scores .85), "at risk" if they were 1 to 2 SD below the mean (scores 70-84), and "delayed" if they were .2SD below the mean (,70). The trajectory of development over time in each domain (cognitive, language, and motor)

SECONDARY OUTCOMES:
neurodevelopment biomarker | intraoperative (before skin incision, end of hypothermia, end of cardiopulmonary bypass), 4 hours after end of surgery
  plasma glial fibrillary acidic protein concentration
inflammation | 4 hours after end of surgery
  level of IL-6
acute kidney injury | 2 hours after end of cardiopulmonary bypass
  urinary NGAL
myocardial injury | intraoperative (before skin incision, end of cardiopulmonary bypass), 4 hours after end of surgery, 24 hours after end of surgery
  level of Troponin i
anesthesia monitoring | intraoperative (from anesthetic induction to end of surgery)
  Bispectral index, end tidal sevoflurane
fluid management | intraoperative (from anesthetic induction to end of surgery)
  amount of transfusion, ROTEM® values
fluid management | intraoperative (from anesthetic induction to end of surgery)
  blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ji SH, Kang P, Song IS, Jang YE, Lee JH, Kim JT, Kim HS, Kim EH. The effect of dexmedetomidine on neuroprotection in pediatric cardiac surgery patients: study protocol for a prospective randomized controlled trial. Trials. 2022 Apr 8;23(1):271. doi: 10.1186/s13063-022-06217-9. PMID 35395776